CLINICAL TRIAL: NCT00266487
Title: Randomized Trial of Homocysteine-lowering With B Vitamins for Secondary Prevention of Cardiovascular Disease After Acute Myocardial Infarction. The Norwegian Vitamin Trial (NORVIT)
Brief Title: The Norwegian Vitamin Trial (NORVIT)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Tromso (Other)
Collaborators: The Research Council of Norway (Other); The Council on Health and Rehabilitation, Norway (Unknown); The Norwegian Council on Cardiovascular Disease (Unknown); The Royal Norwegian Ministry of Health (Other); The International Federation of Red Cross and Red Crescent Societies (Other); Foundation to Promote Research into Functional Vitamin B12 Deficiency, Bergen, Norway (Other)
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: NRC 112812/320; NRC 138859/320
Record Dates: First submitted 2005-12-15; First posted 2005-12-16 (Estimated); Last update posted 2017-05-08 (Actual); Status verified 2017-05

CONDITIONS: Acute Myocardial Infarction
Keywords: Homocysteine; B vitamins; Folic acid; Randomized trial; Secondary prevention
MeSH Terms: interventions — Folic Acid; Vitamin B 12; Vitamin B 6

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Folic acid
Drug: Vitamin B12
Drug: Vitamin B6

SUMMARY:
The purpose of this study is to examine whether the lowering of blood homocysteine levels by treatment with B vitamins can prevent cardiovascular disease

DETAILED DESCRIPTION:
Observational studies have demonstrated that elevated levels of plasma total homocysteine is a risk factor for cardiovascular disease. The purpose of this trial is to evaluate the efficacy of homocysteine lowering treatment with B vitamins for secondary prevention in patients who have experienced an acute myocardial infarction.

This controlled, double-blind, multi-centre trial will include 3750 men and women aged 30-85 who have experienced an acute myocardial infarction within 7 days prior to randomization. Participants will be randomized, in a two-by-two factorial design, to receive one of the following four treatments: A, folic acid 0.8 mg plus vitamin B12 0.4 mg and vitamin B6 40 mg per day; B, folic acid 0.8 mg plus vitamin B12 0.4 mg per day; C, vitamin B6 40 mg per day; D, placebo.

The primary end point during 3.5 years of follow-up is a composite of recurrent myocardial infarction and stroke and sudden death attributed to coronary artery disease.

ELIGIBILITY:
Inclusion Criteria:

* Acute myocardial infarction within 7 days prior to randomization
* Men and women aged 30-85 years
* Written informed consent

Exclusion Criteria:

* Coexisting disease that shortens expected survival to less than 4 years
* Ongoing treatment with B vitamins
* Expected poor compliance

Ages: 30 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3750
Dates: Start 1998-12; Study Completion 2004-03

PRIMARY OUTCOMES:
The primary end point was a composite of
nonfatal myocardial infarction,
fatal myocardial infarction,
nonfatal stroke,
fatal stroke, and
sudden death attributed to coronary heart disease.

SECONDARY OUTCOMES:
Individual components of the primary end point, i.e.
Nonfatal myocardial infarction
Fatal myocardial infarction
Nonfatal stroke
Fatal stroke
In addition the following secondary outcomes:
Unstable angina pectoris requiring hospitalization
Percutaneous coronary revascularization
Coronary-artery bypass grafting
Death from any cause
Cancer
Pulmonary embolus
Transitoric ischemic attack
Surgery for abdominal aortic aneurysm
Plasma homocysteine levels
Plasma levels of B vitamins

CONTACTS AND LOCATIONS:
Overall Officials: Kaare H Bonaa, M.D., Ph.D, Principal Investigator — Institute of Community Medicine, University of Tromsø, Norway
Locations (1):
- Institute of Community Medicine, University of Tromsø, Tromsø, Norway

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Bonaa KH, Njolstad I, Ueland PM, Schirmer H, Tverdal A, Steigen T, Wang H, Nordrehaug JE, Arnesen E, Rasmussen K; NORVIT Trial Investigators. Homocysteine lowering and cardiovascular events after acute myocardial infarction. N Engl J Med. 2006 Apr 13;354(15):1578-88. doi: 10.1056/NEJMoa055227. Epub 2006 Mar 12. PMID 16531614
- [Derived] Dhar I, Lysne V, Svingen GFT, Ueland PM, Gregory JF, Bonaa KH, Nygard OK. Elevated plasma cystathionine is associated with increased risk of mortality among patients with suspected or established coronary heart disease. Am J Clin Nutr. 2019 Jun 1;109(6):1546-1554. doi: 10.1093/ajcn/nqy391. PMID 31005968